CLINICAL TRIAL: NCT03425955
Title: Aesthetic Performance of an Intradermal Injection Treatment for Face Photoaging: Interstitial or Cushion Technique in Comparison to Bolus Technique at Five Points (Half - Face Method Within Subjects)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1817
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Face Photoaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Experimental): Normotypic or overweight subjects with rounded, oval or squared face (aged 35-50 years)
  Interventions: Device: SUNEKOS ® 200
- GROUP 2 (Experimental): Thin subjects with oval or triangular face and "sagging" skin (aged 45-60 years)
  Interventions: Device: "SUNEKOS® 1200" and "SUNEKOS® 200"

INTERVENTIONS:
Device: SUNEKOS ® 200 — 4 micro-injection sessions of "SUNEKOS® 200" with an interval of 10 days. Two different injection techniques were carried out mono-laterally on the left or right face side randomly: "interstitial fluid technique" (IFT) on one face side; bolus technique on five pre-determined face points (zygomatic protuberance, nostril's angle, inferior margin of tragus, lip marionette lines, mandibular angle) on the contralateral face side.
  Arms: GROUP 1
Device: "SUNEKOS® 1200" and "SUNEKOS® 200" — 5 micro-injection sessions (one of the product "SUNEKOS® 1200" and four of "SUNEKOS® 200". "SUNEKOS® 1200" was injected bi-laterally on the face with cushion technique. 24 hours after the "SUNEKOS® 1200" treatment, 4 micro-injection sessions of "SUNEKOS® 200" with an interval of 10 days were performed . "SUNEKOS® 200" was injected with two different techniques, carried out mono-laterally on the left or right face side randomly: "retrograde interstitial fluid technique" (RIFT) on one face side; bolus technique on five pre-determined face points (zygomatic protuberance, nostril's angle, inferior margin of tragus, lip marionette lines, mandibular angle) on the contralateral face side.
  Arms: GROUP 2

SUMMARY:
Aesthetic performance of "SUNEKOS® 200" injectable treatment on main sign of face skin aging in normotypic or overweight subjects with rounded, oval or squared face and in thin subjects with oval or triangular face and "sagging" skin.Interstitial or cushion technique in comparison to bolus technique at five points (half - face method within subjects).

DETAILED DESCRIPTION:
Spontaneous, open, clinical trial, conducted by one centre under dermatological control. Primary end point of the study was to evaluate clinically and by non-invasive instrumental measurements the aesthetic performance of "SUNEKOS® 200" injectable treatment on main sign of face skin aging in normotypic or overweight subjects with rounded, oval or squared face and in thin subjects with oval or triangular face and "sagging" skin.

The micro-injections of the study product were executed by a specialized dermatologist, on the face of female volunteers with photoaging of mild/moderate grade; to improve the treatment aesthetic performance two different injection techniques were carried out mono-laterally on the left or right face side randomly: "interstitial fluid technique" (IFT) for the 1st subjects' typology (aged 35-50 years) and "cushion technique" in association to "retrograde interstitial fluid technique" (RIFT) for the 2nd (aged 45-60). On the contralateral face side the injection treatment was performed by bolus technique on five pre-determined face points, preceding for the 2nd subjects' typology by cushion technique.

It was also aim of this study to evaluate tolerance both by investigator and volunteers and efficacy by the volunteers

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* age 35-50 years for the group 1 and 45-60 years for the group 2,
* mild/moderate cutaneous photoaging according to a reference photographic scale
* skin phototype I, II and III according to Fitzpatrick's classification, with a preference to grade II-III ,
* agreeing to present at each study visit without make-up,
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products,
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study,
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy,
* lactation,
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study,
* subjects not in menopause who do not accept to perform the pregnancy test during the basal visit, 30 days (T4i) and 60 days (T60) after the first injection procedure,
* Body Mass Index (BMI) variation (± 1) during the study period,
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 12 months prior to the study start;
* performing permanent filler in the past,
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test,
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit),
* subjects whose insufficient adhesion to the study protocol is foreseeable,
* presence of cutaneous disease on the tested area, as lesions, scars, malformations,
* recurrent facial/labial herpes,
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* diabetes,
* endocrine disease,
* hepatic disorder,
* renal disorder,
* cardiac disorder,
* pulmonary disease,
* cancer,
* neurological or psychological disease,
* inflammatory/immunosuppressive disease,
* drug allergy,
* anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion. The use of other drugs, not mentioned above, can be authorized by the Investigator.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Variation of wrinkles grade of the area around the eyes | Baseline (T0), immediately after the 1st "Sunekos® 200" injection treatment (T1i), 60 days (T60).
  Reduction of grade of the area around the eyes corresponding to a decrease from the baseline of the Glogau's reference photographic scale clinical score where:
  Type 1 (No Wrinkles) Early photo-aging, mild pigment changes, minimal wrinkles, no 'age spots'; Type 2 (Wrinkles in Motion) Early to moderate photo-aging, appearance of lines only when face moves, early brown 'age spots', skin pores more prominent, early changes in skin texture; Type 3 (Wrinkles at Rest) Advanced photo-aging, prominent brown pigmentation, visible brown 'age spots', prominent and small blood vessels, wrinkles now present with face at rest; Type 4 (Only Wrinkles) Severe photoaging, wrinkles everywhere (at rest or moving) yellow-grey skin color, prior skin cancers, pre-cancerous skin changes (actinic keratosis).
Variation of Wrinkle Severity Rating Scale (WSRS) grade | Baseline (T0), immediately after the 1st "Sunekos® 200" injection treatment (T1i), 60 days (T60).
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  Grade 1 (absent): no visible nasolabial fold; continuous skin line. Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.
Variation of Facial Volume Loss Scale (FVLS) grade | Baseline (T0), immediately after the 1st "Sunekos® 200" injection treatment (T1i), 60 days (T60).
  Reduction of face volume loss corresponding to a decrease from the baseline of the Facial Volume Loss Scale (FVLS) where:
  Grade 1 Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). No prominent bony landmarks. No visibility of underlying musculature.
  Grade 2 An intermediate point between grade 1 and grade 3. Grade 3 Moderate concavity of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas. Prominence of bony landmarks. May have visibility of underlying musculature.
  Grade 4 An intermediate point between grade 3 and grade 5. Grade 5 Severe indentation of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). Severe prominence of bony landmarks. Clear visibility of underlying musculature

SECONDARY OUTCOMES:
Photographic documentation (3D pictures) | Baseline (T0), immediately after the 1st "Sunekos® 200" injection treatment (T1i), 60 days (T60).
  Three-dimensional pictures of the face taken by VECTRA H1 handheld imaging system
Face volume variation | Baseline (T0), immediately after the 1st "Sunekos® 200" injection treatment (T1i), 60 days (T60).
  Face volume image analysis was carried on the 3D pictures taken by Vectra H1 thanks to Vectra analysis module (VAM) software

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy